CLINICAL TRIAL: NCT07017205
Title: Automated Versus Manual Cuff Pressure Control for Preventing Microaspiration With TaperGuard Endotracheal Tubes in Elective Surgery: A Randomized Controlled Trial
Brief Title: Microaspiration and Endotracheal Tubes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Argentinian Intensive Care Society (Other)
Responsible Party: Principal Investigator, Gustavo Plotnikow, Head of Physical and Respiratory Care Department, ICU, HOSPITAL BRITANICO DE BUENOS AIRES
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: PRIISABA15678
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Endotracheal Tube Cuff; Microaspiration; Endotracheal Tube Cuff Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: In addition to the participants, both the investigator responsible for patient randomization and the evaluator analyzing the samples for microaspiration will be blinded to group allocation. This double-masking approach is intended to minimize bias in both the allocation process and the outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Conventional Cuff Pressure Control Group (Active Comparator): Patients will be intubated by experienced anesthesiologists using a TaperGuard Evac tube (Covidien) with tapered cuff and subglottic suction system. Cuff inflation will be performed using the standard method commonly employed in clinical practice (passive recoil of syringe plunger).
  Interventions: Device: Application of oropharyngeal dye and tracheal aspirate collection
- Continuous Cuff Pressure Control Group (Experimental): The intervention group will receive a TaperGuard Evac tube (Covidien) with tapered cuff and subglottic suction system, plus continuous cuff pressure monitoring using the Pressure Easy® device (Medtronic) to maintain 25-30 cmH₂O.
  Interventions: Device: Application of oropharyngeal dye and tracheal aspirate collection

INTERVENTIONS:
Device: Application of oropharyngeal dye and tracheal aspirate collection — After intubation, 2 mL of blue dye will be applied to the oropharyngeal mucosa. Once hemodynamically stable (MAP >65 mmHg), the first tracheal aspirate will be collected within 10 minutes by a blinded investigator for analysis.

SUMMARY:
The goal of this clinical trial is to learn if a new method for managing breathing tube pressure is better at preventing fluid from leaking into patients' lungs during surgery. It will also check if it causes fewer side effects like a sore throat.

The main questions it aims to answer are:

Does using a continuous pressure controller reduce fluid leakage past the breathing tube cuff compared to the standard manual method? Does the continuous pressure controller lead to fewer and less severe sore throats and voice changes after surgery?

Researchers will compare two groups:

Group 1: Patients whose breathing tube cuff pressure is managed with a continuous automatic controller.

Group 2: Patients whose breathing tube cuff pressure is managed with the standard manual method.

Participants will:

Be randomly assigned to one of the two groups before their surgery. Receive a small, safe amount of blue dye in their mouth during the procedure to help measure leakage.

Have two small secretion samples collected from their breathing tube during surgery.

Be asked about sore throat and voice changes at 1, 2, 3, and 24 hours after the breathing tube is removed.

DETAILED DESCRIPTION:
1. The Clinical Challenge: Microaspiration and the Breathing Tube

   Endotracheal intubation is a life-saving procedure, but it inherently bypasses the body's natural defenses against lung infection. A critical, yet often overlooked, problem is microaspiration. This is the silent leakage of small amounts of oropharyngeal secretions past the cuff of the breathing tube and into the lower airways and lungs. This phenomenon is a primary contributor to the development of Ventilator-Associated Pneumonia (VAP), a serious complication that increases patient morbidity, mortality, and healthcare costs.

   The cuff's primary role is to create a seal within the trachea. However, conventional cylindrical cuffs can form folds or channels when inflated, creating a direct pathway for secretions to leak through. Furthermore, maintaining the correct cuff pressure (recommended 25-30 cmH₂O) is challenging; pressure can fluctuate due to patient movement, changes in anesthesia gas volume, and surgical positioning.
2. Technological Innovations and the Evidence Gap

   To address these issues, manufacturers have developed advanced endotracheal tubes. This study focuses on the TaperGuard™ Evac tube (Covidien/Medtronic), which features a uniquely shaped tapered cuff. This design is intended to inflate more uniformly against the tracheal wall, theoretically reducing the formation of leakage channels compared to traditional cylindrical cuffs.

   Concurrently, technology for pressure management has evolved. While the current standard of care involves intermittent manual checks with a manometer, automated cuff pressure controllers (like the Pressure Easy® device) have been introduced. These devices continuously monitor and adjust the pressure, maintaining it within a pre-set target range throughout the entire procedure without manual intervention.

   While laboratory (bench-top) studies strongly suggest that tapered cuffs are superior at preventing fluid leakage, and some early clinical studies are promising, there is a lack of robust, in-vivo evidence from a controlled surgical setting. This study aims to fill that gap by directly testing the combined effect of the advanced tube design with two different levels of pressure management sophistication.
3. The Study's Core Investigation: A Two-Factor Comparison

   This trial is not just testing a new device, but rather investigating a clinical management strategy. The central question is: Does moving from a manual, intermittent pressure management protocol to a continuous, automated one provide a significant clinical benefit when using a modern, tapered-cuff endotracheal tube?

   To answer this, we are employing a rigorous model to objectively quantify microaspiration:

   The Blue Dye Model: A small, safe volume of blue dye is instilled into the patient's oropharynx above the cuff after intubation. The presence or absence of this dye in tracheal aspirate samples, collected later from below the cuff, serves as an objective, binary measure (Yes/No) of whether leakage has occurred.
4. Broader Impact and Secondary Patient-Centered Outcomes

   Beyond the primary goal of preventing pneumonia, the study also investigates patient comfort and safety post-operatively. Damage to the tracheal mucosa from improper cuff pressure or physical irritation from the tube can lead to:

   Post-extubation sore throat: A common and uncomfortable complaint.

   Post-extubation dysphonia: Hoarseness or voice changes resulting from vocal cord irritation.

   By ensuring more stable and optimal cuff pressure, the continuous controller may mitigate these issues. We will track these outcomes using standardized, validated scales (a Numeric Rating Scale for pain and the GRBAS scale for voice quality) to determine if the intervention leads to a tangible improvement in the patient's immediate recovery experience.
5. Methodological Rigor

To ensure the results are reliable and unbiased, the study employs key methodological safeguards:

Randomization: Patients are randomly assigned to a study group using a computer-generated sequence to ensure groups are comparable.

Partial Blinding: While the clinical team at the bedside cannot be blinded to the monitoring device, the laboratory analysis of the tracheal secretion samples is performed by personnel who are completely unaware of which group the sample came from. This prevents bias in determining the primary outcome.

In summary, this study seeks to provide high-quality evidence to guide clinical practice in operating rooms, determining if an investment in automated pressure control technology yields measurable benefits in patient safety and comfort when using state-of-the-art endotracheal tubes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old) scheduled for surgery lasting at least one hour.
* ASA I-III classification.
* Signed informed consent.

Exclusion Criteria:

* Pre-existing airway pathology (e.g., tracheomalacia, granulomas, stenosis, tumors).
* Anticipated difficult intubation (Macocha Score > 3 points).
* Selective lung ventilation / one-lung ventilation.
* Current participation in another clinical trial.

Elimination Criteria:

* Accidental extubation.
* Cardiorespiratory arrest or death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Penetration of blue-dyed oropharyngeal secretions into the distal airway | From enrollment to the end of Surgery: Tracheal aspirate samples will be collected at two defined time points: the first between 10 and 30 minutes after intubation and hemodynamic stabilization, and the second immediately prior to extubation.
  Evaluate the penetration of blue-dyed oropharyngeal secretions into the distal airway in patients undergoing orotracheal intubation.

SECONDARY OUTCOMES:
Real-time changes in endotracheal tube cuff pressure during the surgical procedure | Intraoperative ( surgical procedure)
  Cuff pressure monitoring will be performed at predefined intervals. In the experimental group, continuous cuff pressure monitoring will be conducted using the Pressure Easy® Cuff Pressure Controller. In the control group, cuff pressure will be manually regulated with a manovacuometer, using the syringe-backflow method to adjust pressure.
Determine the incidence of post-extubation pain. | The pain will be assessed at the following post-extubation time points: 1 hour, 2 hours, 3 hours, and 24 hours.
  Post extubation pain evaluated using the verbal numerical rating scale (0-10).
Determine the incidence of post-extubation dysphonia. | These dysphonia will be assessed at the following post-extubation time points: 1 hour, 2 hours, 3 hours, and 24 hours.
  Post-extubation dysphonia: Assessed using the GRBAS (Grade, Roughness, Breathiness, Asthenia, Strain) clinical scale, with the grade aspect scored from 0 to 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Britanico de Buenos Aires, CABA, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dullenkopf A, Gerber A, Weiss M. Fluid leakage past tracheal tube cuffs: evaluation of the new Microcuff endotracheal tube. Intensive Care Med. 2003 Oct;29(10):1849-53. doi: 10.1007/s00134-003-1933-6. Epub 2003 Aug 16. PMID 12923620
- [Background] Lorente L, Lecuona M, Jimenez A, Lorenzo L, Roca I, Cabrera J, Llanos C, Mora ML. Continuous endotracheal tube cuff pressure control system protects against ventilator-associated pneumonia. Crit Care. 2014 Apr 21;18(2):R77. doi: 10.1186/cc13837. PMID 24751286
- [Background] Blot SI, Poelaert J, Kollef M. How to avoid microaspiration? A key element for the prevention of ventilator-associated pneumonia in intubated ICU patients. BMC Infect Dis. 2014 Nov 28;14:119. doi: 10.1186/1471-2334-14-119. PMID 25430629